CLINICAL TRIAL: NCT01328561
Title: The Role of Oxytocin and Arginine Vasopressin in Human Placebo Analgesia
Brief Title: Oxytocin and Arginine Vasopressin in Pain Relief
Status: Terminated | Type: Observational
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 110104; 11-M-0104
Record Dates: First submitted 2011-04-01; First posted 2011-04-04 (Estimated); Last update posted 2018-07-05 (Actual); Status verified 2015-03-04

CONDITIONS: Placebo Analgesia
Keywords: Arginine; Oxytocin; Vasopressin; Placebo; Analgesia; Healthy Volunteer; HV
MeSH Terms: conditions — Diabetes Insipidus; Agnosia

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Background:

- Oxytocin, a substance produced mostly in the brain, plays a role in influencing social interactions and reactions to stress, and may be related to pain. Arginine vasopressin, a hormone that regulates water, sugar, and salt in the blood, influences hostile behaviors and reactions to stress, and may also be related to pain. Researchers are interested in investigating both substances and their relationship to pain in healthy volunteers.

Objectives:

- To evaluate the effects of oxytocin and arginine vasopressin on pain in healthy volunteers.

Eligibility:

- Healthy volunteers between 18 and 55 years of age.

Design:

* This study involves two 2-hour testing sessions held 1 day apart. Each session includes the administration of oxytocin, arginine vasopressin, or placebo (a nonactive substance), or no drug. The drugs and the placebo will be given by a nasal spray.
* At the first visit, participants will provide blood and saliva samples to measure hormone levels, and will be asked to fill out questionnaires about some psychological factors such as anxiety and empathy. Participants will then have an assessment of their sensitivity to pain, consisting of a brief electrical stimulation that lasts less than 1 second. After the pain assessment, participants will receive oxytocin, arginine vasopressin, placebo, or no drug at all, and will be monitored to provide baseline information. Participants will then have another pain sensitivity test and will complete the questionnaires again, and provide another saliva sample.
* At the second visit, participants will provide another saliva sample; receive oxytocin, arginine vasopressin, placebo, or no drug at all; and have tests of pain sensitivity and a pain-relieving procedure. During the pain-relieving procedure, participants will receive brief, moderately painful electrical shocks on the back of the nondominant hand and a low-level electrical stimulation on the middle finger that counteracts or reduces the pain from the shocks. Participants will rate their pain perception at the end of each stimulation by using a visual scale ranging from 0 (no pain) to 10 (maximum imaginable pain). The experiment ends with a final saliva collection and completion of the psychological questionnaires.

DETAILED DESCRIPTION:
Objective:

It is well known that social and contextual cues and the whole atmosphere around the patient, such as words, attitudes, and providers behaviors, all contribute to evoke placebo responses. Moreover, an extensive literature investigating prosocial behaviors (e.g. ability to share another s feelings, imitation, mimicry) suggests that social modeling is critical in developing learning processes across species, including social influences on psychophysical aspects of pain. Only recently, it has been demonstrated that observing the beneficial effects in a demonstrator induces substantial placebo analgesic responses which are positively correlated with empathy. A crucial role in social behaviors is played by oxytocin (OXT) and arginine vasopressin (AVP), two neuropeptides, produced mostly in the hypothalamus and acting on certain brain regions whose function is associated with emotion perception (amygdale and nucleus accumbens), eye-gaze, trust and processing of positive and negative social cues. Since beliefs, trust and contextual cues are important elements of the clinicianpatient relationship and socially-induced placebo effects, it is reasonable to hypothesize that OXT and AVP may be one of the endogenous substances that trigger contextual and interpersonal placebo responses. By viewing interpersonal healing as a central causal process (or a set of related causal processes) within the domain of pain modulation, it is possible to probe the potential role for OXT and AVP in the modulation of a placebo response. In pursuit of this goal, we use a neuropharmacological intervention with OXT and AVP agonists in combination with a behavioral, brain imaging and genetic approach.

Study population:

Healthy men and women participants aging from 18 to 55 years.

Design:

We will investigate the role of oxytocinergic system in the processing of social cues by using a model of pain and interpersonal placebo analgesia already tested (9). The following drugs will be used: 1) oxytocin, 2) arginine vasopressin, and 3) placebo.

Outcome measures:

Primary outcomes are subjective pain reports (Experiment 1) and brain- and cortical -related responses (Experiments 2 and 3). Secondary measures include skin conductance response, heart rate, cortisol, subjective measures of empathy; trait and state anxiety measures; and functional pain-related genetic polymorphisms.

ELIGIBILITY:
* INCLUSION CRITERIA
* Men and Women
* Aged between 18-55 years
* Able to understand and speak the English language

EXCLUSION CRITERIA

* Any significant medical or neurological problems (e.g. cardiovascular illness, respiratory illness, neurologic illness, seizures, etc.)
* History of angioedema
* High blood pressure (above 140 mmHg) or symptomatic low blood pressure
* History of fainting
* A family history of mania, schizophrenia, or other psychoses (first-degree relatives only)
* A history of mania, schizophrenia, or other psychoses
* Any current Axis I psychiatric disorders (e.g. depression and anxiety)
* Lifetime alcohol/drug dependence
* Alcohol/drug abuse in the past year
* Current use of psychotropic medication
* Impaired hearing
* Pregnancy
* Breast-feeding
* Smokers (use of any form of nicotine during the last six months)
* Color-blindness (e.g. difficulty to distinguish between red and green colors)

History of fainting and symptomatic hypotension will be reviewed by the clinicians responsible for the screening and study on a case-by-case basis.

ADDITIONAL EXCLUSION CRITERIA FOR THE MRI AND MEG STUDIES

Participants taking part in the MRI (Experiment 2) and MEG (Experiment 3) studies will also be excluded in case of:

* Metal slivers or shavings lodged in the tissues of the head or neck
* Surgical clips or shrapnel in or near the brain or blood vessels
* Any metallic objects in the eyes or central nervous system, and any form of implant wire or metal device that may concentrate radiofrequency fields
* Head trauma with loss of consciousness in the last year or any evidence of functional impairment due to and persisting after head trauma.
* Previously worked in metal fields or machines that may have left any metallic fragments in or near your eyes.
* Tattooed makeup (eyeliner, lip, etc) or general tattoos in a dangerous location on your body.
* Any non-organic implant or any other device such as: cardiac pacemaker, insulin infusion pump, implanted drug infusion device, cochlear, otologic, or ear implant, transdermal medication patch (Nitro), any metallic implants or objects, body piercing(s), bone/joint pin, screw, nail, plate, wire sutures or surgical staples, or shunt.
* Any psychological contraindications for MRI (e.g., fear of closed places).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 167 (Actual)
Dates: Start 2011-03-17; Study Completion 2015-03-04

CONTACTS AND LOCATIONS:
Overall Officials: Luana Colloca, M.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Colloca L, Benedetti F. Placebos and painkillers: is mind as real as matter? Nat Rev Neurosci. 2005 Jul;6(7):545-52. doi: 10.1038/nrn1705. PMID 15995725
- [Background] Colloca L, Benedetti F, Porro CA. Experimental designs and brain mapping approaches for studying the placebo analgesic effect. Eur J Appl Physiol. 2008 Mar;102(4):371-80. doi: 10.1007/s00421-007-0593-6. Epub 2007 Oct 25. PMID 17960416
- [Background] Zubieta JK, Stohler CS. Neurobiological mechanisms of placebo responses. Ann N Y Acad Sci. 2009 Mar;1156:198-210. doi: 10.1111/j.1749-6632.2009.04424.x. PMID 19338509
- [Derived] Colloca L, Schenk LA, Nathan DE, Robinson OJ, Grillon C. When Expectancies Are Violated: A Functional Magnetic Resonance Imaging Study. Clin Pharmacol Ther. 2019 Dec;106(6):1246-1252. doi: 10.1002/cpt.1587. Epub 2019 Sep 10. PMID 31350784
- [Derived] Colloca L, Grillon C. Understanding placebo and nocebo responses for pain management. Curr Pain Headache Rep. 2014 Jun;18(6):419. doi: 10.1007/s11916-014-0419-2. PMID 24771206